CLINICAL TRIAL: NCT00166504
Title: A Multicenter, Randomized, Open-label Study to Evaluate the Lipid-Altering Efficacy and Safety of Ezetimibe (+) Simvastatin Versus Atorvastatin in Patients With Primary Hypercholesterolemia
Brief Title: Ezetimibe Plus (+) Simvastatin Versus Atorvastatin Comparative Study (0653A-092)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-092; MK0653A-092; 2005_070
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2008-11-05 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vytorin (Experimental): Ezetimibe 10 mg/Simvastatin 20 mg
  Interventions: Drug: ezetimibe (+) simvastatin
- Atorvastatin (Active Comparator): Atorvastatin 10 mg
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — simvastatin/ezetimibe 10/20 mg
  Other Names: MK0653A; Vytorin®
  Arms: Vytorin
Drug: atorvastatin — atorvastatin 10 mg
  Other Names: Lipitor®
  Arms: Atorvastatin

SUMMARY:
This is an efficacy and safety study of Vytorin (ezetimibe (+) simvastatin) compared to atorvastatin (ezetimibe/simvastatin) at week 6 in primary hypercholesterolemia patients in Korea. The primary hypothesis being tested is that daily administration of Vytorin will result in a greater reduction of low density lipoprotein cholesterol (LDL-C) concentration from baseline after 6 weeks treatment compared to atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypercholesterolemia
* LDL-C >/= 130 mg/dL but </=250 mg/dL and triglyceride (TG) </= 350 mg/dL
* National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) III guideline

Exclusion Criteria:

* Hypersensitivity to 3-hydroxy-3-methyl-glutaryl-CoA reductase (HMG-CoA reductase) inhibitors or Ezetimibe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a 4-week diet/wash-out period, patients still at or above drug treatment thresholds established by National Cholesterol Education Program Adult Treatment Panel III Guidelines were randomized. Randomization was stratified according to LDL-C levels obtained 1 week pre-randomization: ≥130 to <160 mg/dL; ≥160 to <190 mg/dL; ≥190 mg/dL.
Period: Overall Study
Arm/Group | Vytorin | Atorvastatin
Started | 108 | 95
Completed | 103 | 91
Not Completed | 5 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vytorin | Atorvastatin | Total
Number analyzed (Participants) | 108 | 95 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.7) | 58.7 (8.7) | 58.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 51 | 39 | 90
Baseline Low Density Lipoprotein Cholesterol (LDL-C) Strata [Number; unit: Participants]
  <130 mg/dl | 2 | 3 | 5
  >=130 to <160 mg/dl | 45 | 32 | 77
  >=160 to <190 mg/dl | 41 | 43 | 84
  >=190 mg/dl | 20 | 17 | 37
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.3 (2.9) | 25 (2.8) | 25.2 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: LDL-C Lowering Efficacy
Description: LDL-C = low density lipoprotein cholesterol, measured in mg/dl.
Time Frame: 6 weeks
Population: Included patients with LDL-C data at both baseline and at the 6-week post-randomization time point.
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Vytorin | Atorvastatin
Number analyzed (Participants) | 105 | 93
Percent Change from Baseline | -51 (14.7) | -41 (16)
Statistical Analysis 1: Comparison: Vytorin vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Net) = -10, 95% CI [-14.3 to -5.7], Standard Deviation 15.3 — Direction of the Comparison: Vytorin minus Atorvastatin

ADVERSE EVENTS:
Arm/Group | Vytorin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/95
Other Adverse Events (participants affected / at risk) | 0/108 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.